CLINICAL TRIAL: NCT02762097
Title: Clinical Pregnancy Rate in Women With Unexplained Infertility After Removal of Unsuspected Intrauterine Pathology
Brief Title: Clinical Pregnancy Rate After Removal of Unsuspected Polyps
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped due to similar case control study already completed
Sponsor: Karachi Medical and Dental College (Other)
Responsible Party: Principal Investigator, samia husain, research assistant, Karachi Medical and Dental College
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: karachiMDC
Record Dates: First submitted 2016-04-30; First posted 2016-05-04 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Infertility
Keywords: polyps; saline sonography; infertility
MeSH Terms: conditions — Infertility; Polyps | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): All women would undergo saline sonography with normal saline. Women with endometrial polyps who consent to the removal of polyps will be offered polypectomy
  Interventions: Procedure: polypectomy; Procedure: saline sonography; Drug: normal saline
- control (Placebo Comparator): All women would undergo saline sonography with normal saline. Women with endometrial polyps who do not consent to the removal would serve as controls
  Interventions: Procedure: saline sonography; Drug: normal saline

INTERVENTIONS:
Procedure: polypectomy — . During the second visit after she consents to removal of polyp revealed on prior saline sonography, a dilatation and curettage would be performed under ultrasound guidance and after successful removal of polyp (polypectomy) saline sonography would be repeated to ensure completeness of removal.
  Arms: intervention
Procedure: saline sonography — saline infusion sonography (SIS) on 8th to 11th day of menstrual cycle. On the day of admission SIS will be performed in an outpatient setting .Taking all aseptic measures a speculum will be inserted vaginally and up to 20 ml of sterile saline solution will be infused into the uterine cavity through a cervical foley's catheter of 5 french to distend the endometrial cavity. A transvaginal transducer will be used to scan the uterine cavity. In case the patient has polyps she would be offered removal under general anaesthesia on a subsequent visit as a day case procedure.
Drug: normal saline — Normal saline would be injected into uterine cavity to delineate defects

SUMMARY:
Polyps are fleshy outgrowths of the inner lining of the womb which may hinder implantation of embryo and lead to subfertility.This study evaluates whether removal of endometrial polyps in womb affects chances of pregnancy in women in whom no other causes of subfertility can be found. Half of the women would have these polyps removed after their consent and the other half who would not consent would not undergo any such intervention

ELIGIBILITY:
Inclusion Criteria:

* Normal semen analysis
* 24 months of unprotected sexual intercourse
* NORMAL TVS
* Normal hysterosalpingogram
* Evidence of spontaneous ovulation
* No history of Pelvic inflammatory disease
* Polyps on saline sonography

Exclusion Criteria:

* History of taking hormones
* Thyroid disorder
* prior hysteroscopy treatment
* intermenstrual blood loss.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-30 (Estimated); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate: | 12 months
  number of women who get pregnancy test positive within 12 months of intervention

IPD SHARING:
Plan to Share IPD: Undecided